CLINICAL TRIAL: NCT06169969
Title: Effect of Magnetic Therapy in Bladder Dysfunction and Quality of Life in Paraplegic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Moataz Mohamed Talaat El Semary, Assistant Professor of physical therapy for neurology and neurosurgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004741
Record Dates: First submitted 2023-11-19; First posted 2023-12-14 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Paraplegia; Spinal Cord Injuries
Keywords: Magnetic therapy; Paraplegia; Bladder dyssynergia; Quality of life
MeSH Terms: conditions — Paraplegia; Spinal Cord Injuries | interventions — Magnetic Field Therapy

STUDY DESIGN:
Intervention Model Description: post hoc test
Who Masked: Participant, Outcomes Assessor
Masking Description: double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnetic therapy group (Experimental): receive magnetic therapy plus pelvic floor exercises.
  Interventions: Device: magnetic therapy
- Pelvic floor exercises group (No Intervention): pelvic floor exercises only

INTERVENTIONS:
Device: magnetic therapy — Kegel exercises
  Other Names: pelvic floor exercises
  Arms: Magnetic therapy group

SUMMARY:
Each study subject will undergo baseline urodynamic testing (UDS) at the beginning of the study to confirm the diagnosis of a neurogenic bladder with DSD and establish baseline bladder functions. The study will be divided into two phases: a Treatment phase (16 weeks) and a Follow-up phase (6 weeks). During the treatment phase, each subject will undergo once/week magnetic spinal cord stimulation (MSCS) at 1Hz (low) frequency (40-60% intensity) over the lumbar spine. Once each subject entered the treatment phase of the study and will receive weekly lumbar spinal cord magnetic stimulation for a total of 16 weeks. This 16-week period of MSCS constituted bladder rehabilitation. Each subject will receive non-video urodynamic testing once every four weeks during the treatment phase to monitor progress and ensure that bladder function will not further impaired. After the initial four-week stimulation period, each subject will be asked to attempt volitional urination for 5-10minutes prior to bladder catheterization. the subjects will instruct to keep the environment quiet, relax and focus on voiding

DETAILED DESCRIPTION:
Forty male Paraplegic patients will be recruited.…from outpatients' clinics and their ages from 20 to 35 years and the inclusion criteria for the study will be a stable American Spinal Injury Association Impairment Scale (AISA) A/B, motor complete spinal cord injury between spinal levels T6-T12 present for greater than 1 year, and a documented history of neurogenic bladder requiring intermittent catheterization. Each subject will require to have at least three prior urodynamic studies to confirm the diagnosis of neurogenic bladder with detrusor sphincter dyssynergia (DSD), which was diagnosed with urodynamic study in which a rise in detrusor pressure and concomitant needle EMG activity and rise in urethral pressure were demonstrated Patients with a history of autonomic dysreflexia were excluded from the study. Any patient who will be ventilator dependent, abusing drugs, have musculoskeletal dysfunction (i.e., unstable fractures), cardiopulmonary diseases, active infections or ongoing depression requiring treatment, or have previous exposure to and use of spinal cord stimulation will be excluded from the study. Patients with a history of bladder Botox injection or bladder/sphincter surgeries will be excluded

ELIGIBILITY:
IInclusion Criteria:

* Male Participants ages 20 to 35 years
* Participants will be a stable American Spinal Injury Association Impairment Scale (AISA) A/B.
* Motor incomplete spinal cord injury between spinal levels T6-T12.
* Participants present for more than 1 year.
* Each participant will require at least three prior urodynamic studies to confirm the diagnosis of neurogenic bladder with detrusor sphincter dyssynergia (DSD), which was diagnosed with urodynamic study.

Exclusion Criteria:

* Patients with a history of autonomic dysreflexia.
* Any patient who will be ventilator dependent, abusing drugs, have musculoskeletal dysfunction (i.e., unstable fractures).
* Any patient who will have cardiopulmonary diseases, active infections or ongoing depression requiring treatment, or have previous exposure to and use of spinal cord stimulation.
* Patients with a history of bladder Botox injection or bladder/sphincter surgeries.

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — ISLAMIC ISSUES
Enrollment: 40 (Actual)
Dates: Start 2023-11-05 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2024-03-04 (Actual)

PRIMARY OUTCOMES:
Bladder Volume at first desire to void in Milliliters. | Baseline, pre-intervention then Peri procedurally after 8 weeks and finally "immediately after the intervention (16 weeks)
  one of bladder functions using urodynamic testing
Detrusor pressure At Qmax in Centimeters of water | Baseline, pre-intervention then Peri procedurally after 8 weeks and finally "immediately after the intervention (16 weeks)
  one of bladder functions using urodynamic testing
Maximum flow rate in milliliters per second | Baseline, pre-intervention then Peri procedurally after 8 weeks and finally "immediately after the intervention (16 weeks)
  one of bladder functions using urodynamic testing
Amplitude per time in millivolts | Baseline, pre-intervention then Peri procedurally after 8 weeks and finally "immediately after the intervention (16 weeks)
  EMG Measurement during contraction of pelvic floor muscles
Upper centile amplitude in millivolts | Baseline, pre-intervention then Peri procedurally after 8 weeks and finally "immediately after the intervention (16 weeks)
  EMG Measurement during contraction of pelvic floor muscles
Qualiveen short version 8 questions from 1 to 4 (worse if high score) | Baseline, pre-intervention then Peri procedurally after 8 weeks and finally "immediately after the intervention (16 weeks)
  Qualiveen questionnaire short form of quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No